CLINICAL TRIAL: NCT06652685
Title: Molecular Subtype Combined with Early Minimal Residual Disease to Optimize the Treatment of Young Treatment-naive Acute Myeloid Leukemia: a Multicenter, Phase II Study
Brief Title: Molecular Subtype Combined with Early Minimal Residual Disease to Optimize the Treatment of Newly Diagnosed Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Shen yang, Vice Director of Hematology Division, Ruijin Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IA+X 2024
Record Dates: First submitted 2024-10-15; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute myeloid leukemia; venetoclax; gilteritinib; D5-PBCR; Risk-stratified
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Subjects receive IA regimen as the initial induction. On day five of induction, D5-PBCR will be tested according to protocol. Patients will be assigned to different arms according to the result of D5-PBCR.
  For FLT3 mutate patients, a combination of gilteritinib will be recommended in this study. Induction and consolidation phase: gilteritinib 80mg on D8-14.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- D5-PBCR(-) (Experimental): On day five of IA induction, D5-PBCR will be tested according to protocol. For D5-PBCR (-) patients, no additional of venetoclax is needed.
  Interventions: Drug: D5-PBCR(-) IA arm
- D5-PBCR(+) (Experimental): On day five of induction, D5-PBCR will be tested according to protocol. D5-PBCR (+) patients, will receive induction therapy consisting of venentoclax combined with IA regimen.
  Interventions: Drug: D5-PBCR(+) IA+Venetoclax arm

INTERVENTIONS:
Drug: D5-PBCR(-) IA arm — Induction: IA Drug: idarubicin, intravenously, 10 mg/m^2 on D1-3 Drug: cytarabine, intravenously, 100 mg/m^2 on D1-7
  Consolidation:
  Subjects who achieve composite complete remission (CRc) proceed with consolidation therapy.
  In consolidation therapy phase, subjects in the group with favorable/intermediate risk and MRD negetive, will receive cytarabine intravenously at 2g/m^2/q12h*6 doses. Subjects in the group with adverse risk or MRD positive will receive cytarabine intravenously at 2g/m^2/q12h*6 doses together with venetoclax 400mg on D4-10. Dose ramp-up of venetoclax is not required.
  After two cycles of consolidation, a multi-disciplinary team will discuss whether the patient need allogeneic hematopoietic stem-cell transplant (allo-HSCT) according to ELN risk stratification and MRD status.
  Arms: D5-PBCR(-)
Drug: D5-PBCR(+) IA+Venetoclax arm — Induction: IA+Ven Drug: idarubicin, intravenously, 10 mg/m^2, on D1-3, Drug: cytarabine, intravenously, 100 mg/m^2 on D1-7 For D5-PBCR (+) patients, Venetoclax will be combined. Drug: Venetoclax. Orally once daily, on D6-14. A 3-day dose ramp-up is required for the first induction (100mg D6, 200mg D7, 400mg D8-14) If a second induction is needed, the dose of IA is the same as the first cycle, and dose ramp-up of venetoclax is not required.
  Consolidation:
  Subjects who achieve composite complete remission (CRc) proceed with consolidation therapy.
  In consolidation therapy phase, subjects in the group will receive cytarabine intravenously at 2g/m^2/q12h*6 doses together with venetoclax 400mg on D4-10. Dose ramp-up of venetoclax is not required.
  After two cycles of consolidation, a multi-disciplinary team will discuss whether the patient need allogeneic hematopoietic stem-cell transplant (allo-HSCT) according to ELN risk stratification and MRD status.
  Arms: D5-PBCR(+)

SUMMARY:
This study aims to investigate the safety and efficacy of drug "X" in combination with intensive chemotherapy in subjects with newly diagnosed AML (excluding APL and CBF-AML). "X" drugs included BCL-2 inhibitor venetoclax and FLT3 inhibitor Gilteritinib.

Subjects will receive standard intensive chemotherapy during induction and consolidation. Early induction response will be evaluated according to the results of peripheral blood blast clearance rate on the fifth day after induction therapy (D5-PBCR). Venetoclax will be added in D5-PBCR positive subjects. For subjects with FLT3 mutations, Gilteritinib will be combined.

Subjects will be stratified based on the genetic risk classification of 2022 European LeukemiaNet recommendations (ELN risk) and MRD status to receive specific consolidation therapy after the induction therapy.

DETAILED DESCRIPTION:
Young patients with naïve AML (excluding APL and CBF-AML) were included in this study. 218 subjects who meet the eligibility criteria will receive the standard 3+7 intensive chemotherapy induction, containing cytarabine and idarubicin. On the basis of the IA induction regimen, the early chemotherapy response was evaluated according to the results of peripheral blood blast clearance rate on the fifth day after induction therapy (D5-PBCR). For D5-PBCR-positive patients, venetoclax will be added to conventional chemotherapy. For patients with FLT3 mutations, gilteritinib will be combined.

Subjects who achieve a composite complete remission (CRc) after induction therapy will receive further consolidation therapy, which regimen will be decided based on the ELN risk at diagnosis and MRD status detected by MFC and gene quantification after induction therapy.

The purpose of the study is to determine whether the addition of drug "X" to the standard induction regimen improves efficacy in the treatment of naïve AML.

Primary objective: To evaluate whether intensive IA combined with targeted drug (drug "X") regimens can improve the composite response rate (CRc) after 1 course of induction therapy in newly diagnosed young AML patients Secondary Objective: To evaluate whether intensive chemotherapy combined with drug "X" during induction and consolidation can improve overall response rates, overall survival, and event-free survival in newly diagnosed young AML patients Safety indicators: incidence of adverse reactions during treatment, recovery time of neutrophils and platelets

ELIGIBILITY:
Inclusion Criteria:

1. Bone marrow morphology and immunology confirmed newly diagnosed AML patients (according to 2022 ICC criteria)
2. Exclude patients with APL and CBF-AML (according to fusion genes and chromosomes)
3. Performance status score 0-2 (ECOG score)
4. Age 18~59 years old
5. Liver and kidney function: blood bilirubin ≤ 35 μmol/L, AST/ALT below 2 times the upper limit of normal, creatinine ≤ 150 μmol/L
6. Normal cardiac function (EF ≥50%)
7. Obtained informed consent signed by the patient or family member

Exclusion Criteria:

1. FAB classification is M3, or confirmed APL at the molecular level
2. CBF-AML
3. Patients who have already been treated
4. Comfirmed central nervous system leukemia
5. Allergy to any of the drugs involved in the protocol
6. Medical condition or organ system dysfunction that precludes the inability to swallow capsules or tablets, or has a disease that significantly affects gastrointestinal function and/or inhibits small bowel absorption (including malabsorption syndrome, small bowel resection, or poorly controlled inflammatory bowel disease)
7. Cardiac function and disease consistent with one of the following: a) long QTc syndrome or QTc interval >480 ms; b) second- or third-degree atrioventricular block; Severe, uncontrolled cardiac arrhythmias requiring medication; c) United States New York College of Cardiology Grade ≥ III; d) Ventricular ejection fraction (LVEF) less than 50%; e) History of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, history of clinically severe pericardial disease, or ECG evidence of acute ischemic or active conduction abnormalities within 6 months prior to recruitment
8. Previous or present concomitant malignancies (except for basal cell carcinoma of the skin that have been effectively controlled as non-melanoma, carcinoma in situ of the breast/cervix, and other malignancies that have not been effectively controlled for more than 6 months, and patients who have been receiving long-term non-chemotherapy treatments such as hormonal therapy)
9. Significant abnormalities in liver and kidney function (serum bilirubin, aspartate aminotransferase, alanine aminotransferase or serum creatinine more than 2 times the upper limit of normal reference values; Excluded from AML-related as judged by the investigator)
10. Patients who have previously used other drugs for the treatment of AML (except hydroxyurea and cytarabine for cell count control), including but not limited to BCL2, FLT3, IDH1, IDH2 inhibitors, or other drugs in clinical trials
11. Coagulopathy not associated with AML
12. HIV infection, syphilis infection, HCV infection, active HBV infection (HBsAg positive, or HBsAg negative but HBcAb positive with HBV DNA > 1.0 ×ULN)
13. Other uncontrolled active infection (as judged by the investigator)
14. Pregnant or lactating women
15. Inability to understand or follow the study protocol
16. Participation in other relevant clinical studies within 30 days (except diagnostic clinical studies)
17. Patients who in the opinion of the investigator, are not suitable to participate in this study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission rate | At the end of cycle one (up to 42 days from the start of cycle 1）
  Complete remission/complete remission with partial hematological recovery/complete remission with incomplete hematological recovery

SECONDARY OUTCOMES:
Total composite complete remission rate | At the end of induction cycle 2 (up to 42 days from the start of cycle 2)
  Complete remission/complete remission with partial hematological recovery/complete remission with incomplete hematological recovery
OS | 2-year
  overall survival rate
EFS | 2-year
  event free survival rate
AE | Throughout the entire study period, an average of 1 year
  Adverse Events (AEs), Serious Adverse Events (SAEs) Based on NCI-CTCAE 5.0 Assessment
Recovery time for neutrophils and platelets | During induction cycle one (up to 42 days from the start of cycle 1)
  The time from the first day of induction therapy to the recovery of neutrophils to a count greater than 0.5*10^9/L and platelets to greater than 20*10^9/L

OTHER OUTCOMES:
The complete remission rate of MRD negative | at the end of induction (up to 42 days from the start of induction cycle 2) and consolidation stage (after two cycles of consolidation, up to 42 days from the start of consolidation cycle 2)
  The complete remission rate of MRD negative
biomarkers of apoptosis | Throughout the entire study period, an average of 1 year
  Level of apoptosis biomarkers such as BCL-2, BCL-xL and MCL-1

CONTACTS AND LOCATIONS:
Overall Officials: Yang Shen, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Li X, Weng X, Shen Y, Chen Y, Zheng Y, Zhao H, You J, Mao Y, Wang L, Wu M, Sheng Y, Wu J, Hu J, Chen Q, Li J. Optimization of idarubicin and cytarabine induction regimen with homoharringtonine for newly diagnosed acute myeloid leukemia patients based on the peripheral blast clearance rate: A single-arm, phase 2 trial (RJ-AML 2014). Am J Hematol. 2022 Jan 1;97(1):43-51. doi: 10.1002/ajh.26386. Epub 2021 Nov 1. PMID 34687467
- [Background] Yu C, Kong QL, Zhang YX, Weng XQ, Wu J, Sheng Y, Jiang CL, Zhu YM, Cao Q, Xiong SM, Li JM, Xi XD, Chen SJ, Chen B. Clinical significance of day 5 peripheral blast clearance rate in the evaluation of early treatment response and prognosis of patients with acute myeloid leukemia. J Hematol Oncol. 2015 May 10;8:48. doi: 10.1186/s13045-015-0145-1. PMID 25957890